CLINICAL TRIAL: NCT01751217
Title: Family Therapy Via Video Teleconference for Substance-Abusing Rural Adolescents
Acronym: RAFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01DA032260-01A1 (NIH)
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Substance-Related Disorders
Keywords: Substance Abuse; Adolescents; Families; Functional Family Therapy; Video; Teleconferencing; Telemedicine
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Funct Family Tx/Video Teleconf (FFT-V) (Experimental): Functional Family Therapy (FFT) is a brief treatment for youth with problem behaviors, including substance abuse that consists of 12 to 14 weekly family sessions. The FFT treatment is applied in five distinct phases: Engagement, Motivation, Relational Assessment, Behavior Change, and Generalization and each phase has specific goals, techniques, and therapist skills. Adolescents and parents assigned to the FFT-V condition will receive a Verizon netbook laptop computer equipped with the Microsoft Windows 7 operating system, webcam, and VTC software for use in the family home. The VTC software is designed to stream live video between therapists and participants, to record video, and to store recorded videos as digital mpeg files. All family sessions will take place via video teleconference.
  Interventions: Behavioral: Functional Family Tx
- Functional Family Tx (Experimental): Functional Family Therapy (FFT) is a brief treatment for youth with problem behaviors, including substance abuse that consists of 12 to 14 weekly family sessions. The FFT treatment is applied in five distinct phases: Engagement, Motivation, Relational Assessment, Behavior Change, and Generalization and each phase has specific goals, techniques, and therapist skills. Families in the FFT condition will not be provided with the laptop and internet access described above. Instead, adolescents and parents in this condition will receive the FFT intervention face-to-face from an FFT therapist who will travel to the family home for each session.
  Interventions: Behavioral: Functional Family Tx
- Services as Usual (Active Comparator): The main CYFD service provider for adjudicated youth in both Sandoval and Valencia counties is Youth Development Incorporated (YDI) which is a private not-for-profit youth service organization serving adolescents in New Mexico . YDI provides an array of services for youth including tutoring, after-school activities, gang intervention, school drop-out prevention, family counseling services, an emergency teen shelter, parenting skills training, youth leadership development, community corrections services, GED studies, substance abuse and AIDS education, etc. The YDI juvenile corrections services include intensive supervision, educational and employment assistance, community service, victim restitution, and institutional transition services.
  Interventions: Behavioral: Services as Usual

INTERVENTIONS:
Behavioral: Functional Family Tx
  Other Names: FFT
  Arms: Funct Family Tx/Video Teleconf (FFT-V); Functional Family Tx
Behavioral: Services as Usual
  Arms: Services as Usual

SUMMARY:
The current proposal is a randomized clinical trial testing the efficacy of Functional Family Therapy (FFT) administered by video teleconference (FFT-V) in the homes of substance abusing adolescents. In the proposed investigation, FFT-V will be compared with FFT administered face-to-face in the family home as well as to a services-as-usual (SAU) condition. The overarching objective of the study is to examine the degree to which an empirically based model of substance abuse treatment such as FFT can be effectively administered via video teleconferencing to adolescents and families living in rural and remote areas who would be otherwise unlikely to access treatment. The specific aims of the proposed study are to (1) evaluate the efficacy of FFT-V compared to FFT and SAU in reducing adolescent drug use, HIV risk behavior, delinquency, and recidivism, (2) evaluate the efficacy of FFT-V compared to FFT in establishing functional levels of therapeutic alliance formation, treatment attendance, retention, and satisfaction with treatment, (3) evaluate the efficacy of FFT-V compared to FFT and SAU in impacting core mechanisms of change in adolescent behavior including improved levels of family functioning and adolescent association with substance using peers, and (4) conduct a preliminary cost-effectiveness analysis to derive initial estimates of the relative costs of each treatment modality per outcome unit.

DETAILED DESCRIPTION:
It has been well documented that only about 10% of adolescents with clinically diagnosable substance use problems receive treatment in any given year. One of the major contributing factors to chronic levels of unmet need for treatment among this population is the unavailability and inaccessibility of treatment services. Service accessibility is particularly limited in rural areas. To address problems of service availability and accessibility in rural areas, the use of video teleconferencing technology to provide direct services has emerged within the fields of medicine and psychiatry in particular. The use of such technology to enhance the delivery of behavioral psychotherapy is beginning to emerge as well. A handful of primarily small-scale pilot and feasibility studies indicate that psychotherapy interventions administered using video teleconferencing technology may be as effective as traditional face-to-face interventions. Few randomized clinical trials of telepsychotherapy have been conducted to date, however, and virtually none have examined video teleconferencing interventions for any type of child or adolescent behavioral problem including substance abuse. The proposed study is intended to address the need for research evaluating the application of video teleconferencing technology as a means of service delivery for substance abusing adolescents and their families living in rural areas. Specifically, this study will examine the efficacy of Functional Family Therapy administered by video teleconference (FFT-V) in the homes of substance abusing adolescents. FFT-V will be compared with FFT administered face-to-face in the family home as well as to services-as-usual (SAU) coordinated through the Juvenile Services Division (JSD) of the State of New Mexico Children, Youth, and Families Department (CYFD). FFT, based on more than 30 years of research, is an established EBT for adolescent substance abuse and related problem behaviors such as HIV risk and delinquency. Moreover, FFT is one of few evidence-based therapies shown to be effective for rural families. The study will be conducted in the homes of participating adolescents and parents living in rural communities located between 30 and 50 miles from the Center for Family and Adolescent Research (CFAR) in Albuquerque, NM. One hundred and twenty youth will be referred to the study by Children Youth and Family Department juvenile probation officers within two rural counties in New Mexico, Sandoval and Valencia, which are adjacent to the town of Albuquerque which is located in Bernalillo County. Adolescent participants meeting diagnostic criteria for substance abuse or dependence, along with the participating parent, will be randomly assigned to the FFT, FFT-V, or SAU conditions. Four assessments of all participants in all three conditions will occur at: pre-treatment, 4-, 8-, and 12 months after treatment initiation. Outcome analyses will examine adolescent substance abuse, HIV risk behavior, delinquency, and recidivism, family functioning, and adolescent association with substance abusing peers. The study will also examine clinical process variables known to impact treatment efficacy (e.g., therapeutic alliance formation, treatment motivation, and retention). The overarching objective of the study is to examine the degree to which an empirically based model of substance abuse treatment such as FFT can be effectively administered via video teleconferencing to adolescents and families living in rural and remote areas and thus have less access to treatment.

ELIGIBILITY:
Inclusion Criteria:

* 13-18 years of age
* Meet DSM-IV diagnostic criteria for substance abuse or dependence
* Reside with at least one parent or parental figure who is willing to participate in the study
* Reside in a rural community approximately 30-50 miles from the CFAR office
* Have sufficient residential stability to permit contact with CFAR throughout the study (e.g., not homeless or runaway at time of intake).

Exclusion Criteria:

* Incarcerated or in a restrictive placement outside the home (e.g., residential treatment, in-patient care)
* Evidence of a psychotic or organic state of sufficient severity to interfere with the ability to understand the research and clinical procedures
* A sibling is already participating in the study
* Evidence of posing a danger to self or others based on routine safety screening protocols (see Intake below)
* Evidence that more intensive services other than outpatient treatment are required (e.g., in-patient care, detoxification).

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2012-02; Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Timeline Followback semi-structured interview (TLFB) | Up to 12-months after randomization
  The TLFB is a semi-structured interview pertaining to substance use behavior over a specific time interval (e.g., past 90 days). On each day of the assessment period, the type and amount of substance use is recorded based on retrospective self-reports. The interviewer utilizes a daily calendar and other types of memory aides to facilitate recall. At the pre-treatment assessment the TLFB will be used to assess the quantity and frequency of adolescent substance use during the 90 days prior to entry into the study. Days spent in a restrictive environment will be excluded from the baseline assessment period. At each post-treatment assessment, the calendar period will extend back to the date of the previous assessment. The TLFB will be used to determine the percent days of substance use excluding tobacco, as well as abstinence days and binge drinking days.

SECONDARY OUTCOMES:
Urine Assays - NIDA 9 Test Panel | up to 12-months after randomization
  The NIDA 9 Test Panel is a card device with 9 finger-like prongs which are dipped in a urine sample to screen for AMP (amphetamine), BAR (barbiturates), BZO (benzodiazepines), COC (cocaine), M-AMP (metamphetamine), MTD (methadone), MOR (morphine), PCP, and THC (marijuana).

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Ozechowski, Ph.D., Principal Investigator — Oregon Research Institute's Center for Family and Adolescent Research; Holly B Waldron, Ph.D, Principal Investigator — Oregon Research Institute's Center for Family and Adolescent Development
Locations (1):
- Oregon Research Institute Center for Family and Adolescent Research, Albuquerque, New Mexico, United States